CLINICAL TRIAL: NCT05524571
Title: A Phase 3, Multi-center, Randomized, Quadruple-masked, Placebo-controlled Study of Batoclimab for the Treatment of Participants With Active Thyroid Eye Disease (TED)
Brief Title: Study to Assess Batoclimab in Participants With Active Thyroid Eye Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMVT-1401-3202
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Eye Disease
Keywords: Batoclimab; Thyroid eye disease; IMVT-1401; Monoclonal antibody; Autoimmune disorders; Graves' Ophthalmopathy; Graves' Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor Staff is also masked, so the study is Quadruple-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Batoclimab (Experimental): Participants will be administered batoclimab 680 mg SC weekly for 12 weeks followed by 340 mg SC weekly for 12 weeks.
  Interventions: Drug: Batoclimab
- Placebo (Placebo Comparator): Participants will be administered matching placebo SC weekly for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Batoclimab — Batoclimab is a fully human anti-neonatal fragment crystallizable receptor (FcRn) monoclonal antibody
  Other Names: IMVT-1401
  Arms: Batoclimab
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of batoclimab 680 milligrams (mg) subcutaneous (SC) once a week (QW) for 12 weeks followed by 340 mg SC QW for 12 weeks versus placebo on proptosis responder rate at Week 24.

ELIGIBILITY:
Inclusion criteria:

1. Are ≥18 years of age at screening.
2. Have a clinical diagnosis of TED associated with active, moderate to severe TED with the following at screening and Visit 0:

   * A CAS ≥ 4 in either eye, and
   * Clinical evidence of worsened proptosis with:

     * Proptosis ≥ 18 mm and/or
     * Proptosis ≥ 3 mm increase from participant's baseline (prior to diagnosis of TED), as estimated by the Investigator/assessor
3. Have moderate to severe active TED, as defined by European Group on Graves' Orbitopathy (EUGOGO) guidelines.
4. Have onset of active TED within 12 months prior to screening.
5. Have documented evidence of detectable anti-TSHR-Ab at screening.
6. Are not expected to require immediate surgical intervention and are not planning corrective surgery/irradiation or medical therapy for TED during the course of the study.
7. Are euthyroid with the Baseline disease under control or have mild hypo- or hyperthyroidism.

Additional inclusion criteria are defined in the protocol.

Exclusion criteria:

1. Have decreased best corrected visual acuity due to optic neuropathy.
2. Have at least a 2-point decrease in CAS or ≥2 mm decrease in proptosis between screening and Baseline assessments in either eye.
3. Have used any steroid (intravenous or oral) for the treatment of TED or other conditions within 4 weeks prior to screening.
4. Have used any steroid (Intravenous or oral) with a cumulative dose equivalent to ≥ 1 g of methylprednisolone for the treatment of TED.
5. Have known autoimmune disease other than TED, that, in the opinion of the Investigator, would interfere with the course and conduct of the study.
6. Had previous orbital irradiation or surgery for TED.

Additional exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of proptosis responders | At Week 24
  Proptosis is the amount of protrusion of the eye from the orbital rim. Measurements are recorded using the Hertel exophthalmometer. The study eye is defined as the most severely affected eye at the Baseline visit. Proptosis responder is defined as the participant with a greater than or equal to (≥) 2 millimeters (mm) reduction in the study eye without deterioration (≥2 mm increase) in the fellow eye.

SECONDARY OUTCOMES:
Percentage of participants with proptosis ≥2 mm reduction and Clinical Activity Score (CAS) of less than or equal to (≤) 3 from Baseline in the study eye | Baseline and Week 24
  The CAS measures the classical signs of acute inflammation (pain, redness, and swelling) in TED. The 7-item scale assigns 1 point for the presence of each of the parameters assessed: spontaneous retrobulbar pain, pain on attempted upward or downward gaze, redness of eyelids, redness of conjunctiva, swelling of caruncle or plica, swelling of eyelids, swelling of conjunctiva (chemosis). The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity. Higher scores indicate worse symptoms.
Percentage of participants with CAS of 0 or 1 in the study eye | At Week 24
Mean change from Baseline in CAS in the study eye | Baseline and Week 24
Percentage of participants with positive binding anti-thyroid stimulating hormone receptor (TSHR) antibody (Ab) at Baseline who achieve seroconversion | Baseline and Week 24
Percentage of participants with decrease of at least 1 grade from Baseline in Gorman score for diplopia | Baseline and Week 24
  Diplopia will be assessed based on 3 grades: Grade I - Intermittent diplopia (diplopia in primary position of gaze, when tired or when first awakening), Grade II - Inconstant diplopia (diplopia at extremes of gaze) and Grade III - Constant diplopia (continuous diplopia in primary or reading position). Higher scores indicate worse symptoms.
Mean change from Baseline in proptosis in the study eye | Baseline and Week 24
Percentage of participants with ≥6-point increase from Baseline in total Graves' ophthalmopathy - Quality of life (GO-QOL) score | Baseline and Week 24
  The GO-QOL is a 16-item self-administered questionnaire designed to assess how GO affects different aspects related to quality of life (visual functioning and psychosocial consequences). The points given to questions 1 to 8 and 9 to 16 are added to obtain 2 raw scores ranging from 8 to 24; one for visual functioning and one for appearance. Higher scores indicate better outcome.
Percentage of participants with ≥8-degree increase from Baseline in motility (in at least 1 of 4 directions) in the study eye | Baseline and Week 24

CONTACTS AND LOCATIONS:
Locations (45):
- United States (15):
  - Site Number -1520, Pasadena, California
  - Site Number -1517, San Francisco, California
  - Site Number -1514, Torrance, California
  - Site Number -1510, Sarasota, Florida
  - Site Number -1516, Louisville, Kentucky
  - Site Number - 1526, Livonia, Michigan
  - Site Number - 1513, Rochester, Minnesota
  - Site Number - 1512, Winston-Salem, North Carolina
  - Site Number - 1525, Portland, Oregon
  - Site Number -1515, Bellaire, Texas
  - Site Number - 1524, McAllen, Texas
  - Site Number -1519, San Antonio, Texas
  - Site Number - 1521, Seattle, Washington
  - Site Number -1511, Morgantown, West Virginia
  - Site Number - 1518, Milwaukee, Wisconsin
- Site Number - 7565, Sydney, Australia
- Belgium (5):
  - Site Number -4671, Bruges
  - Site Number - 4672, Brussels
  - Site Number - 4673, Brussels
  - Site Number -4670, Ghent
  - Site Number - 4674, Liège
- Site Number - 6603, Mainz, Rhineland-Palatinate, Germany
- Hungary (3):
  - Site Number - 7550, Budapest
  - Site Number - 7551, Pécs
  - Site Number - 7552, Pécs
- Latvia (3):
  - Site Number -9301, Ogre
  - Site Number -9300, Riga
  - Site Number - 9302, Ventspils
- New Zealand (2):
  - Site Number - 7570, Christchurch
  - Site Number - 7572, Hamilton
- Site Number -1990, San Juan, Puerto Rico
- Slovakia (4):
  - Site Number - 9203, Bratislava
  - Site Number - 9200, Bratislava
  - Site Number - 9201, Bratislava
  - Site Number - 9202, Trenčín
- Spain (7):
  - Site Number -3602, Barcelona
  - Site Number - 3605, Barcelona
  - Site Number -3601, Madrid
  - Site Number -3604, Madrid
  - Site Number -3600, Santiago de Compostela
  - Site Number -3606, Seville
  - Site Number -3603, Valencia
- Turkey (Türkiye) (3):
  - Site Number - 4952, Adana
  - Site Number - 4950, Ankara
  - Site Number - 4951, Istanbul

IPD SHARING:
Plan to Share IPD: No